CLINICAL TRIAL: NCT03472963
Title: Body Compartment Pharmacokinetics of Anti-retroviral Agents That May be Used for Future HIV Post-exposure Prophylaxis Regimens.
Brief Title: Body Compartment Pharmacokinetics of Anti- Retroviral Agents That May be Used for Future HIV Post- Exposure Prophylaxis.
Acronym: PEP2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colleen Kelley, Associate Professor, Emory University
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: IRB00101179
Record Dates: First submitted 2018-03-15; First posted 2018-03-21 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: HIV Infections
Keywords: Post-Exposure Prophylaxis; Anti-Retroviral; Pharmacokinetics
MeSH Terms: conditions — HIV Infections | interventions — Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (8):
- Pre- drug (No Intervention): Participants will not receive any drug. They will be asked to return 1-6 weeks after the screening visit for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, rectal swabs, urine sample, and rectal biopsy via rigid sigmoidoscopy.
- Group A.1 (Experimental): Men will be dosed with Genvoya and Darunavir® on site (time of dose will be recorded) and asked to return in 2 hours, 24 hours (+/- 1 hour), and 72 hours (+/- 1 hour) after taking dose for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, and a urine sample). Participant will undergo rectal swabs and rectal biopsy via rigid sigmoidoscopy in 2 hours after dosing.
  Interventions: Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir®
- Group A.2 (Experimental): Men will be dosed with Genvoya and Darunavir® on site (time of dose will be recorded) and asked to return in 2 hours, 24 hours (+/- 1 hour), and 72 hours (+/- 1 hour) after taking dose for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, and a urine sample). Participant will undergo rectal swabs and rectal biopsy via rigid sigmoidoscopy in 24 hours after dosing.
  Interventions: Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir®
- Group A.3 (Experimental): Men will be dosed with Genvoya and Darunavir® on site (time of dose will be recorded) and asked to return in 2 hours, 24 hours (+/- 1 hour), and 72 hours (+/- 1 hour) after taking dose for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, and a urine sample). Participant will undergo rectal swabs and rectal biopsy via rigid sigmoidoscopy in 72 hours after dosing.
  Interventions: Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir®
- Group B.1 (Experimental): Men will be dosed with Genvoya and Darunavir® on site (time of dose will be recorded) and asked to return in 4 hours, 48 hours (+/- 1 hour), and 96 hours (+/- 1 hour) after taking dose for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, and a urine sample). Participant will undergo rectal swabs and rectal biopsy via rigid sigmoidoscopy in 4 hours after dosing.
  Interventions: Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir®
- Group B.2 (Experimental): Men will be dosed with Genvoya and Darunavir® on site (time of dose will be recorded) and asked to return in 4 hours, 48 hours (+/- 1 hour), and 96 hours (+/- 1 hour) after taking dose for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, and a urine sample). Participant will undergo rectal swabs and rectal biopsy via rigid sigmoidoscopy in 48 hours after dosing.
  Interventions: Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir®
- Group B.3 (Experimental): Men will be dosed with Genvoya and Darunavir® on site (time of dose will be recorded) and asked to return in 4 hours, 48 hours (+/- 1 hour), and 96 hours (+/- 1 hour) after taking dose for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, and a urine sample). Participant will undergo rectal swabs and rectal biopsy via rigid sigmoidoscopy in 96 hours after dosing.
  Interventions: Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir®
- Group C (Experimental): Participants will be given a one- day supply of with Genvoya and Darunavir®. Participants return 8 hours (+/- 30min window), 24 hours (+/- 1 hr), and 48 hours (+/- 1 hour) after taking dose for study procedures (blood collection, oral cheek swab, penile swabs, urethral swab, and a urine sample). Participant will undergo rectal swabs and rectal biopsy via rigid sigmoidoscopy in 8 hours after taking the medication.
  Interventions: Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir®

INTERVENTIONS:
Drug: Single dose of Genvoya® and a single 800 mg dose of Darunavir® — Men will be instructed to take Single dose of Genvoya® and a single 800 mg dose of Darunavir® per oral
  Arms: Group A.1; Group A.2; Group A.3; Group B.1; Group B.2; Group B.3; Group C

SUMMARY:
This study is being conducted to determine if the uptake of anti-HIV medications called Genvoya® and darunavir is different at several body sites, including mucosal tissues.

DETAILED DESCRIPTION:
Men who have sex with men (MSM) continue to be disproportionately affected by HIV. The majority of MSM acquire HIV after exposure to the rectal mucosa through unprotected receptive anal intercourse. Post-exposure-prophylaxis (PEP) is an intervention that is used to prevent HIV infection soon (72 hours) after a potential exposure. HIV-negative people with a possible exposure to HIV are instructed to take 28 days of a combination anti-HIV medication regimen, Truvada® + Raltegravir. This study is being conducted to determine if the uptake of other anti-HIV medications called Genvoya® and darunavir is different at several body sites, including mucosal tissues. These other medications might be considered for PEP regimens in the future.

ELIGIBILITY:
Inclusion Criteria:

1. HIV-negative man who reports receptive anal sex with another man in the last 6 months
2. Aged 18-49 years
3. Not currently taking PrEP and no plans to initiate during study
4. Not currently taking PEP
5. Able to provide informed consent in English
6. No plans for relocation in the next 3 months
7. Willing to undergo peripheral blood, penile swabs, urine, and rectal biopsy sampling
8. Willing to use study products as directed
9. Willing to abstain from receptive anal intercourse 3 days prior to starting study product and for the duration of the study and for 7 days after any rectal biopsy procedure.

Exclusion Criteria:

1. History of inflammatory bowel disease or other inflammatory, infiltrative, infectious or vascular condition involving the lower gastrointestinal tract that, in the judgment of the investigators, may be worsened by study procedures or may significantly distort the anatomy of the distal large bowel
2. Significant laboratory abnormalities at baseline visit, including but not limited to:

   1. Hgb ≤ 10 g/dL
   2. PTT > 1.5x ULN or INR > 1.5x ULN
   3. Platelet count <100,000
   4. Creatinine clearance <60
3. Any known medical condition that, in the judgment of the investigators, increases the risk of local or systemic complications of endoscopic procedures or pelvic examination, including but not limited to:

   1. Uncontrolled or severe cardiac arrhythmia
   2. Recent major abdominal, cardiothoracic, or neurological surgery
   3. History of uncontrolled bleeding diathesis
   4. History of colonic, rectal, or vaginal perforation, fistula, or malignancy
   5. History or evidence on clinical examination of ulcerative, suppurative, or proliferative lesions of the anorectal mucosa, or untreated sexually transmitted disease with mucosal involvement
4. Continued need for, or use during the 14 days prior to enrollment, of the following medications:

   1. Aspirin or more than 4 doses of NSAIDs
   2. Warfarin, heparin (low-molecular weight or unfractionated), platelet aggregation inhibitors, or fibrinolytic agents
   3. Any form of rectally administered agent besides lubricants or douching used for sexual intercourse
5. Continued need for, or use during the 90 days prior to enrollment, of the following medications:

   1. Systemic immunomodulatory agents
   2. Supraphysiologic doses of steroids
   3. Experimental medications, vaccines, or biologicals
6. Intent to use HIV antiretroviral pre/post-exposure prophylaxis (PrEP or PEP) during the study, outside of the study procedures
7. Symptoms of an untreated rectal sexually transmitted infection (e.g. rectal pain, discharge, bleeding, etc.)
8. Current use of hormonal therapy
9. Any other clinical condition or prior therapy that, in the opinion of the investigator, would make the patient unsuitable for the study or unable to comply with the study requirements.

Ages: 18 Years to 49 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 35 (Actual)
Dates: Start 2018-04-27 (Actual); Primary Completion 2019-03-29 (Actual); Study Completion 2019-03-29 (Actual)

PRIMARY OUTCOMES:
Median Genvoya plasma concentration | 2 to up to 96 hours after time of dose
  Approximately 24 mL of blood will be drawn to obtain Genvoya plasma concentration (median + range; ng/mL)
Median Darunavir plasma concentration | 2 to up to 96 hours after time of dose
  Approximately 24 mL of blood will be drawn to obtain Darunavir plasma concentration (median + range; ng/mL)
Median Genvoya rectal tissue distribution | 2 to up to 96 hours after time of dose
  Rectal biopsy via rigid sigmoidoscopy will be performed to obtain Genvoya rectal tissue distribution (median + range; ng/mg of tissue).
Median Darunavir rectal tissue distribution | 2 to up to 96 hours after time of dose
  Rectal biopsy via rigid sigmoidoscopy will be performed to obtain Darunavir rectal tissue distribution (median + range; ng/mg of tissue).

SECONDARY OUTCOMES:
Median Genvoya rectal secretion concentration | 2 to up to 96 hours after time of dose
  Rectal swabs for Genvoya rectal secretion concentration (median + range; ng/swab)
Median Darunavir rectal secretion concentration | 2 to up to 96 hours after time of dose
  Rectal swabs for Darunavir rectal secretion concentration (median + range; ng/swab)
Median Genvoya urethral secretion concentration | 2 to up to 96 hours after time of dose
  Urethral swab for Genvoya urethral secretion concentration (median + range; ng/swab)
Median Darunavir urethral secretion concentration | 2 to up to 96 hours after time of dose
  Urethral swab for Darunavir urethral secretion concentration (median + range; ng/swab)

CONTACTS AND LOCATIONS:
Overall Officials: Colleen Kelley, MD, MPH, Principal Investigator — Emory University
Locations (1):
- Emory University, Atlanta, Georgia, United States